CLINICAL TRIAL: NCT04200339
Title: Adolescent SCreening To Help Eliminate Misuse
Acronym: ASC-THEM
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry); Friends Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Sharon Levy, Director, Adolescent Substance Use and Addiction Program, Boston Children's Hospital
Other Study IDs: CTN0060-A1; UG1DA015831 (NIH)
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Substance Use
Keywords: Screening; Adolecents; SBIRT; Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents: Adolescents between the ages of 12 and 17 years old (inclusive).

SUMMARY:
The specific aim of this study is to evaluate the performance of three substance use screening instruments (S2BI, BSTAD, and TAPS Tool) against a criterion standard of Diagnostic Statistical Manual - 5 (DSM-5) substance use disorder (SUD) diagnoses in an adolescent population.

DETAILED DESCRIPTION:
This study seeks to evaluate the psychometric properties of three substance use screening and brief assessment tools for adolescents against criterion standard of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) substance use disorder diagnoses in a population of adolescents who receives care at a participating primary care practice; or, for an initial evaluation at a substance use disorders program for youth. The three tools to be tested are the Brief Screener for Tobacco, Alcohol and Drugs (BSTAD); Screening to Brief Intervention (S2BI) screening tool; and the Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool. BSTAD and S2BI were developed specifically for use with adolescents and each has been validated in a single trial. These tools use past-year "frequency of use" questions to determine risk level for a substance use disorder. The TAPS tool includes both screening and brief assessments and while it has been studied more extensively in adult primary care patients, its validity with adolescents is not known. For youth, alcohol, marijuana and tobacco use, and particularly early initiation, are associated with greater risk of substance use disorders, use of illicit drugs, misuse of opioids, and opioid use disorders. Thus, identifying and addressing substance use early is an important form of prevention that can be delivered in medical care settings for this age group.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 12-17 years, inclusive, at the time of screening.
2. A patient registered at one of the primary care sites; or, presenting for an initial substance use disorders evaluation at the youth substance use disorders program site.
3. Be willing and able to participate in the study.

Exclusion Criteria:

1. Previously enrolled in the current study, as determined by the Chart Review Log/Clinical Staff Referral Log and through self-report of potentially eligible participants.
2. Inability to comprehend spoken or written English.
3. Inability to self-administer any type of computer tool due to physical limitations.
4. Physical or emotional illness that interferes with participation on the day of the appointment, as determined by either the clinical team or research team.
5. Per participant self-report, treated in a residential/inpatient substance use disorders treatment program within the past 12 months.
6. For patients at primary care sites, current, self-reported enrollment in a substance use disorders treatment program at time of recruitment.
7. Per participant self-report, participant is currently in the custody of the Department of Youth Services, the Department of Children and Families, or living with a foster family.
8. Per participant self-report, currently pregnant or parenting.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Recruitment and study procedures may occur either in-person or remotely. We will recruit participants to enroll in the study from participating health care sites. These will include 1) an outpatient adolescent substance use disorders program at a pediatric hospital (ASAP, Boston Children's Hospital), 2) the adolescent medicine program at a federally qualified health center (FQHC) in Boston (Martha Elliot Health Center (MEHC), Boston Children's Hospital), and 3) community-based primary care pediatrics practices that participate in the Pediatric Physicians' Organization at Children's (PPOC). The FQHC is considered a primary care sites participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
SUD assessment evaluation for performance | single visit
  The focus of this study is to evaluate the performance of each tool (S2BI, BSTAD, and TAPS Tool) in identifying substance use and substance use disorders at previously identified cut points for alcohol, marijuana and tobacco/nicotine for each tool. The properties that will be evaluated include sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (LR+) and negative likelihood ratio (LR-)
SUD assessment evaluation for criterion measures | single visit
  We will examine each substance from each tool against the corresponding substance on the criterion standard measure. For example, the tobacco item on the BSTAD would be compared to the tobacco item on the WMH CIDI.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens Hopsital - Adolecents Substance Use and Addiction Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Implementation Guidance(https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm). Investigators will also register and report results of the trial in ClinicalTrials.gov, consistent with the requirements of the Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration (https://grants.nih.gov/policy/clinical-trials/reporting/understanding/nih-policy.htm).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: upon completion
Access Criteria: Public:
  Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the NIDA Data Share Agreement.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Derived] Levy S, Minegishi M, Brogna M, Subramaniam G, McCormack J, Weiss R, Weitzman ER. Comparing the Performance of World Mental Health Composite International Diagnostic Interview Substance Abuse Module in Adolescents to Diagnoses Made by Pediatric Addiction Medicine Specialists. J Addict Med. 2024 Mar-Apr 01;18(2):205-208. doi: 10.1097/ADM.0000000000001271. Epub 2024 Jan 30. PMID 38289239